CLINICAL TRIAL: NCT06425926
Title: A Phase 1/2, Open-label, Multi-center Study of the Safety, Tolerability, and Efficacy of GIM-531 as a Single Agent and in Combination With Anti-PD-1 in Advanced Solid Tumors
Brief Title: Safety and Tolerability Study of GIM-531 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Georgiamune Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GIM531-CT01
Record Dates: First submitted 2024-05-16; First posted 2024-05-23 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Melanoma Stage IV; Solid Tumor
Keywords: PD-1 resistance; PD-1 resistant/refractory; AKT3
MeSH Terms: conditions — Melanoma | interventions — spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 Single Agent (Experimental): GIM-531 administered orally daily
  Interventions: Drug: GIM-531
- Phase 2 Combination Treatment (Experimental): GIM-531 administered orally daily in combination with anti-PD-1 therapy
  Interventions: Drug: GIM-531; Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Drug: GIM-531 — GIM-531 administered orally daily
Drug: Anti-PD-1 monoclonal antibody — Continued treatment with anti-PD-1 therapy
  Arms: Phase 2 Combination Treatment

SUMMARY:
GIM-531 is a first-in-class, orally bioavailable small molecule that is being developed for the treatment of advanced solid tumors as a single agent and rescue therapy. GIM-531 exhibits its primary effect through selective inhibition of regulatory T-cells (Tregs).

DETAILED DESCRIPTION:
GIM531-CT01 is a Phase 1/2 open label, first-in-human, multicenter study. The Phase 1 portion will include a dose escalation with GIM-531 administered as a single agent. Additionally, there will be a dose expansion portion at the safety-cleared dose levels with participants allocated 1:1 within the proposed therapeutic range to accrue additional data for determining the safety profile, pharmacokinetics (PK) profile, pharmacodynamic (PD) effects and early anti-tumor activity of GIM-531. In Phase 2, GIM-531will be administered to participants with advanced/metastatic cutaneous melanoma who have progressed following treatment with an anti-PD-1 therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent
* Cytologically or histologically confirmed locally advanced or metastatic solid tumor that has progressed on standard therapy or for which no standard therapy exist; or be intolerant of standard therapy
* Have not received an experimental drug within 4 weeks or 5 half-lives (whichever is shorter) of study drug treatment or already be enrolled in a clinical study
* ECOG performance status 0-1
* Laboratory and ECG assessments within 28 days of enrollment including acceptable cardiac, renal, and hepatic functions
* Agree to baseline core needle biopsy or archival (within 12 months of screening) tumor submission; Note: Participants whose only site(s) of disease are in areas considered moderate or high risk for biopsy complications may be enrolled without a fresh biopsy upon Sponsor approval.
* Non pregnant participants; female participants of child bearing potential with non-sterile partners agree to use an effective form of contraception from the time of first dose of study drug (or 14 days prior to first dose for oral contraception) until 7 months after the last dose of study drug. Effective forms of contraception include hormonal (injection or oral), double barrier method, or intrauterine device. Non-sterile male participants with sexual partners of childbearing potential agree to use a barrier contraception method and agree to not donate sperm from the time of first dose of study drug until 4 months after the last dose of study drug.
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1

Phase 1 Expansion Cohorts Specific Inclusion Criteria (in addition to above inclusion criteria):

* NSCLC: Participants must have locally advanced/unresectable or metastatic NSCLC. Participants must have received no more than 3 prior lines of therapy in the advanced/metastatic setting.
* TNBC: Participants must have locally advanced unresectable, recurrent, or metastatic TNBC. Participants must have received no more than 3 prior lines of therapy in the advanced/metastatic setting.
* Ovarian Cancer: Participants must have locally advanced unresectable, recurrent, or metastatic ovarian cancer. Participants must have platinum-resistant ovarian cancer defined as disease recurrence or within 6 months after the last administration of platinum-based chemotherapy. Participants must have received no more than 1 line of therapy after development of platinum resistance. Maintenance treatment with Poly(ADP-ribose) polymerase inhibitors (PARPi) or bevacizumab are not counted as separate lines of therapy.
* Tumors with AKT3 mutation/amplification: Participants must have a locally advanced unresectable, recurrent, or metastatic solid malignancy. Participants with known AKT3 mutation/amplification based on next generation sequencing (NGS) performed per local standard of care.

Phase 2 Specific Inclusion Criteria (in addition to above inclusion criteria):

* Have confirmed unresectable Stage III or metastatic Stage IV cutaneous melanoma, NSCLC, or RCC that has radiographically progressed (as confirmed by imaging assessed by the Investigator) on an approved single-agent or combination anti-PD-1 therapy
* Must have received the anti-PD-1 therapy containing regimen as the latest line of treatment and be eligible to restart or to continue anti-PD-1 therapy in combination with GIM-531
* BRAF wild-type melanoma or RCC: Participants must have received no more than 2 prior lines of therapy in the advanced/metastatic setting
* BRAF (V600) mutant melanoma or NSCLC: Participants must have received no more than 3 prior lines of therapy in the advanced/metastatic setting.

Key Exclusion Criteria:

* Ongoing >Grade 1 toxicity from prior therapy according to Common Terminology Criteria for Adverse Events v5.0 (Note: Grade 2 alopecia and Grade 2 sensory neuropathy are not exclusionary)
* Has known leptomeningeal disease, spinal cord compression, or brain metastases, except participants with the following:

  * Brain metastases that have been treated and are clinically stable for at least 4 weeks prior to the first administration of study drug; Note: Participants receiving steroids for brain metastases must be either off steroids or on a stable, or decreasing dose, of <10 mg daily of prednisone (or equivalent) in order to be eligible for enrollment; and
  * No ongoing neurological symptoms related to the anatomic location of the brain metastases.

Note: Neurological symptoms that are considered sequelae to treatment for brain metastases are allowed.

* Has known structural cardiac disease
* Has known serious arrythmia, serious dysrhythmia, history of long QT syndrome, or clinically relevant cardiac conduction abnormalities
* Has an active autoimmune disease that has required systemic treatment in the past 12 months (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* At time of screening, is receiving systemic steroid therapy (greater than or equal to 10 mg/day of prednisone or equivalent) or is taking any immunosuppressive therapy; Note: Use of topical, inhaled, nasal, or ophthalmic steroids is allowed.
* Has active and clinically significant bacterial, fungal, or viral infection, including known hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
* Has a history of, or currently has, an acquired or primary (congenital) immunodeficiency;
* Has had prior anti-cancer treatment with chemotherapeutic agents or immune modulating agents within <4 weeks or 5 half-lives, whichever is shorter, prior to the first dose of study drug.
* Has received a live vaccine within 30 days of first dose of study drug;
* Has had or has planned major surgery within 2 weeks of the first dose of study drug;
* Inability to swallow an oral dose of a medication (eg, oral capsules)
* Is taking medications that are considered strong inducers or inhibitors of CYP2C8 or CYP3A4/5, P-glycoprotein (P-gp), breast cancer resistant protein (BCRP), or sensitive substrates of P-gp and BCRP (Appendix C) that cannot be discontinued at least 1 week prior to first dose of study drug and for the duration of the study.
* Is taking drugs that modify gastric pH, such as proton-pump inhibitors (PPIs) or H2 blockers. Antacids such as calcium carbonate or aluminum hydroxide-based products are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) / serious adverse events (SAEs) and tolerability | Through study completion, an average of 1 year
  To assess incidence and severity of AE / SAEs and tolerability assessed by CTCAE grading
Dose limiting toxicities (DLT) with GIM-531 | 21 days
  To identify dose limiting toxicities with GIM-531

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Predose, 0.5, 1, 2, 4, 6, 8, 24 hours post-dose
  To preliminarily evaluate the Cmax in patients with advanced solid tumors
Time to maximum plasma concentration (Tmax) | Predose, 0.5, 1, 2, 4, 6, 8, 24 hours post-dose
  To preliminarily evaluate Tmax in patients with advanced solid tumors
Area under the plasma concentration versus time curve (AUC) | Predose, 0.5, 1, 2, 4, 6, 8, 24 hours post-dose
  To preliminarily evaluate the AUC in patients with advanced solid tumors
Objective response rate (ORR) | From study enrollment until participant discontinuation, first occurrence of progressive disease, or death from any cause, whichever occurs first (approximately 2 years)
  To identify objective response rate in patients with advanced solid tumors
Best overall response (BOR) | From study enrollment until participant discontinuation, first occurrence of progressive disease, or death from any cause, whichever occurs first (approximately 2 years)
  To preliminarily evaluate BOR in patients with advanced solid tumors
Duration of response (DOR) | From study enrollment until participant discontinuation, first occurrence of progressive disease, or death from any cause, whichever occurs first (approximately 2 years)
  To preliminarily evaluate DOR in patients with advanced solid tumors
Disease control rate (DCR) | From study enrollment until participant discontinuation, first occurrence of progressive disease, or death from any cause, whichever occurs first (approximately 2 years)
  To preliminarily evaluate DCR in patients with advanced solid tumors
Progression-free survival (PFS) | From study enrollment until participant discontinuation, first occurrence of progressive disease, or death from any cause, whichever occurs first (approximately 2 years)
  To preliminarily evaluate PFS in patients with advanced solid tumors
Overall survival (OS) rates | From study enrollment until death from any cause (OS rate assessed at 12 months)
  To preliminarily evaluate OS in patients with advanced solid tumors, including 12 month OS
Tumor expression of immunological markers | Cycle 1 Days 1, 2 and 8; Cycle 2 Days 1 and 8; Cycle 3 Day 1 (each Cycle is 14 days)
  To analyze tumor expression of immunological markers

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Providence Medical Foundation, Fullerton, California
  - The Angeles Clinic and Research Institute, A Cedars-Sinai Affiliate, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Intermountain Health St. Vincent Regional Hospital - Cancer Centers of Montana, Billings, Montana
  - Weill Cornell Medicine - New York Presbyterian Hospital, New York, New York
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No